CLINICAL TRIAL: NCT02216773
Title: Liver Regeneration: a Single-centre, Prospective, Randomised Controlled Trial Comparing Radiofrequency Assisted Liver Partition With Portal Vein Ligation (RALPP) With Portal Vein Embolization (PVE) for Preoperative Induction of Liver Hypertrophy in Patients With Insufficient Future Liver Remnant Volume for Major Liver Resection.
Brief Title: Regeneration of Liver: Portal Vein Embolization Versus Radiofrequency Assisted Ligation for Liver Hypertrophy (REBIRTH)
Acronym: REBIRTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14/LO/1123
Record Dates: First submitted 2014-08-05; First posted 2014-08-15 (Estimated); Results first posted 2019-11-07 (Actual); Last update posted 2019-11-07 (Actual); Status verified 2019-10

CONDITIONS: Liver Resection; Cancer
Keywords: Liver hypertrophy; Liver resection; Liver metastases; Portal vein ligation; Portal vein embolization; Radiofrequency splitting
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Portal vein embolization (PVE) (Active Comparator): Patients allocated to the PVE group will receive pre-intervention blood tests and a contrast enhanced CT scan of the abdomen. They will then have their portal vein embolized radiologically once their pre-intervention investigations have been completed and reviewed by the clinical team.
  Post-intervention investigations (blood tests and CT scan) will take place 4 weeks after the completion of the PVE. At this point, they will be listed to receive their definitive surgical hepatectomy.
  Interventions: Procedure: Portal vein embolization (PVE)
- Radiofrequency assisted liver partition and ligation (RALPP) (Experimental): Patients allocated to the RALPP group will receive pre-intervention blood tests and a contrast enhanced CT scan of the abdomen. They will then have their right portal vein surgically ligated followed by radiofrequency ablation in situ splitting of the liver. Certain patients may additionally have a tumourectomy or wedge resection of the left liver lobe if clinically indicated. The RALPP procedure will occur once the patient's pre-intervention investigations have been completed and reviewed by the clinical team.
  Post-intervention investigations (blood tests and CT scan) will take place 2 weeks after the completion of the RALPP. At this point, they will be listed to receive their definitive surgical hepatectomy.
  Interventions: Procedure: Radiofrequency assisted liver partition with portal vein ligation (RALPP)

INTERVENTIONS:
Procedure: Radiofrequency assisted liver partition with portal vein ligation (RALPP)
  Arms: Radiofrequency assisted liver partition and ligation (RALPP)
Procedure: Portal vein embolization (PVE)
  Arms: Portal vein embolization (PVE)

SUMMARY:
The aim of this study is to compare two different techniques (portal vein embolization and radiofrequency assisted liver partition with portal vein ligation) for increasing liver volume prior to major liver resection.

DETAILED DESCRIPTION:
Liver resection remains the gold standard treatment for patients with liver tumours providing them the only chance for long-term survival. In up to 45% of cases that are amenable to surgical resection, an extended hepatectomy (removal of part of the liver) is usually necessary to achieve a clear resection margin. However, there must be enough liver left behind to meet the demands of the body. Indeed, liver failure due to insufficient remnant liver volume is still the principal cause of postoperative death following a major liver resection.

The liver receives its main blood supply from two vessels (the portal vein and the hepatic artery). In order to decrease the complications and improve the safety of extensive liver surgery in patients with insufficient future liver remnant volume (FLRV), pre-operative embolization (i.e. blockage) of part of the portal vein can be undertaken.

This has the effect of inducing growth of the liver on the unaffected side. Thus, when the resection is carried out, an increased FLRV (of around 12%) reduces post-operative liver failure. An alternative technique is to perform surgical ligation of the portal vein along with splitting of the liver.

The diseased portion of liver is left in the body for 7-10 days while the healthy side is induced to grow. During this time, the diseased portion continues to support the body's requirement for liver function and reduces the risk of liver failure. FLRV has been shown to increase by around 74% with this technique.

However, there are more postoperative complications with the alternative technique such as bile leaks. The aim of this study is to test a new way of splitting the liver so that the increased FLRV can be achieved without the increased complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Any patient requiring right or extended right hepatectomy with FLRV less than 25% on preoperative volumetric study
* WHO performance status 0, 1 or 2
* Patient able to comply with protocol requirements and deemed fit for surgical resection
* Written informed consent

Exclusion Criteria:

* Inability to give informed consent
* Pregnancy
* WHO status 3 or 4
* New York Heart Association Classification Grade III or IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Long R Jiao, MD, FRCS, Principal Investigator — Imperial College London
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gall TM, Sodergren MH, Frampton AE, Fan R, Spalding DR, Habib NA, Pai M, Jackson JE, Tait P, Jiao LR. Radio-frequency-assisted Liver Partition with Portal vein ligation (RALPP) for liver regeneration. Ann Surg. 2015 Feb;261(2):e45-6. doi: 10.1097/SLA.0000000000000607. No abstract available. PMID 24670841

RESULTS

PARTICIPANT FLOW:
Groups:
- Portal Vein Embolization (PVE): Patients allocated to the PVE group received pre-intervention blood tests and a contrast enhanced CT scan of the abdomen. They then had their portal vein embolized radiologically once their pre-intervention investigations were completed and reviewed by the clinical team.
  Post-intervention investigations (blood tests and CT scan) occurred 4 weeks after the completion of the PVE. At this point, they were listed to receive their definitive surgical hepatectomy.
  Portal vein embolization (PVE)
- Radiofrequency Assisted Liver Partition and Ligation (RALPPS): Patients allocated to the RALPP received pre-intervention blood tests and a contrast enhanced CT scan of the abdomen. They then had their right portal vein surgically ligated followed by radiofrequency ablation in situ splitting of the liver. Certain patients may also have had a tumourectomy or wedge resection of the left liver lobe if clinically indicated. The RALPPS procedure occurred once the patient's pre-intervention investigations were completed and reviewed by the clinical team.
  Post-intervention investigations (blood tests and CT scan) occurred 2 weeks after the completion of the RALPPS. At that point, they were listed to receive their definitive surgical hepatectomy.
  Radiofrequency assisted liver partition with portal vein ligation (RALPPS)
Period: Overall Study
Arm/Group | Portal Vein Embolization (PVE) | Radiofrequency Assisted Liver Partition and Ligation (RALPPS)
Started | 28 | 29
Underwent Procedure (PVE/RALPPS) | 24 | 26
Completed | 16 | 24
Not Completed | 12 | 5
Not completed — Disease progression | 4 | 2
Not completed — Insufficient FLRV | 4 | 0
Not completed — Abandoned | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Portal Vein Embolization (PVE) | Radiofrequency Assisted Liver Partition and Ligation (RALPPS) | Total
Number analyzed (Participants) | 24 | 26 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (8.9) | 62.4 (10.2) | 63.3 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 12 | 15 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Changes in Liver Remnant Volume
Description: Percentage change in remnant liver volume following intervention. This will be measured by volumetric analysis of CT scan. Positive number represents increases and negative number represents decreases.
Time Frame: 2 or 4 weeks post intervention (2 weeks post RALPP; 4 weeks post PVE)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Portal Vein Embolization (PVE) | Radiofrequency Assisted Liver Partition and Ligation (RALPPS)
Number analyzed (Participants) | 24 | 26
percentage change | 18.4 (9.8) | 80.7 (13.7)

2. Secondary Outcome: Postoperative Liver Function Tests
Description: Blood tests
Time Frame: Postoperatively (daily until discharge; then at clinic appointments up to 18 months from randomization)
Population: Data not collected
Arm/Group | Portal Vein Embolization (PVE) | Radiofrequency Assisted Liver Partition and Ligation (RALPPS)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Postoperative Complications (Dindo Clavien ≥Grade 3b)
Description: As defined by Dindo Clavien classification of surgical complications (≥grade 3b).
Time Frame: Up to hospital discharge (estimated to be between 2 and 10 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Portal Vein Embolization (PVE) | Radiofrequency Assisted Liver Partition and Ligation (RALPPS)
Number analyzed (Participants) | 24 | 26
Participants | 1 | 4

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Portal Vein Embolization (PVE) | Radiofrequency Assisted Liver Partition and Ligation (RALPPS)
All-Cause Mortality (participants affected / at risk) | 0/24 | 1/26
Serious Adverse Events (participants affected / at risk) | 1/24 | 4/26
Other Adverse Events (participants affected / at risk) | 13/24 | 10/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Portal Vein Embolization (PVE) (N=24) | Radiofrequency Assisted Liver Partition and Ligation (RALPPS) (N=26)
Postoperative complication (Dindo Clavien ≥grade 3b) (Surgical and medical procedures) | 1 (1) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Portal Vein Embolization (PVE) (N=24) | Radiofrequency Assisted Liver Partition and Ligation (RALPPS) (N=26)
Postoperative complication (Dindo Clavien <grade 3b) (Surgical and medical procedures) | 13 (13) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT02216773/Prot_SAP_000.pdf